CLINICAL TRIAL: NCT04451031
Title: Evaluation of the Impact of Linking Families and Teens (LiFT) Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philliber Research & Evaluation (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sally Brown, Senior Research Associate, Philliber Research & Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00017127
Record Dates: First submitted 2020-06-19; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LiFT Program (Experimental): LiFT is a two-module curriculum workshop for youth and their parenting adults. Topics for youth include communication skills, condom use, and skill building to access sexual healthcare resources. For parenting adults, topics include building a climate of trust and open communication with youth about sexual health. Trained and certified facilitators deliver each 2.5 hour module over one or two sessions. Youth and parents participated in simultaneous but separate programming in community locations such as schools or health care settings. They received participant guides that encourage communication between them. They could opt-in to receive 12 weekly texts that offered additional resources. Parenting adults received a phone call from the facilitator a month after the workshop to reinforce the skills learned during the program.
  Interventions: Behavioral: LiFT Program
- Comparison Group (No Intervention): The comparison group received business as usual. The youth and parents enrolled in the study could receive the existing services available within the broader community, which may have included sexual education delivered in the local school system. Study staff collected data throughout the study to track access to other TPP programming offered at the study sites.

INTERVENTIONS:
Behavioral: LiFT Program
  Arms: LiFT Program

SUMMARY:
To test a new curriculum designed by Planned Parenthood of the Great Northwest and Hawaiian Islands (PPGNHI). The Linking Families and teens (LiFT) curriculum is an innovative program designed for families in rural communities, with the goal of reducing unplanned teen pregnancies by increasing family connectedness and increasing youth's self-efficacy, knowledge, and skills related to sexual health.

DETAILED DESCRIPTION:
LiFT is a two-module curriculum workshop for youth and their parenting adults. Topics for youth include communication skills, condom use, and skill building to access sexual healthcare resources. For parenting adults, topics include building a climate of trust and open communication with youth about sexual health.

Trained and certified facilitators delivered each 2.5 hour module. Sites could choose to deliver the modules in one or two sessions. Youth and parents participated in simultaneous but separate programming in community locations such as schools or health care settings. Youth and parenting adults also received participant guides that encouraged communication between them. Facilitators encouraged youth and parenting adults to opt-in to receive weekly texts that offer additional resources and suggestions for fun ways families can communicate; these continued for 12 weeks after the workshop. Parenting adults received a phone call from the facilitator 3 to 5 weeks after the workshop to reinforce the skills learned during the program.

Community partners (schools, health care settings, or other community organizations) assisted with recruiting interested dyads of youth and parenting adults from their client base and the community. Each site held a kickoff event or individual meeting or meetings describing the LiFT program in detail.

Over the course of three years, the program was offered 57 times across five cohorts. The program took place in rural communities across nine states; Alaska, California, Hawaii, Idaho, Mississippi, New York, Oregon, Utah, and Washington. The study enrolled 886 dyads for participation.

The LiFT study was a cluster randomized controlled trial. Dyads of youth and their parenting adults were randomly assigned to participate in the intervention or comparison group. Siblings were randomly assigned together within the same condition. At kick-off events or through individual meetings, program staff obtained parental consent and student assent and administered baseline surveys. After receiving consent, assent, and baseline surveys, the research team conducted the random assignment of dyads and informed the site of the results. Program implementation occurred within two weeks of recruitment and baseline data collection.

All study participants were surveyed at two points in time: (1) at the kickoff event or individual meetings before random assignment (baseline) and (2) immediately post-program (3 months from baseline). In addition, youth were surveyed 1 year following baseline. LiFT facilitators administered the baseline surveys, whereas the evaluation team administered the immediate post-program and 9-month post-program follow-up surveys. Surveys were in-person pencil-and-paper surveys for all survey points. Dyads who did not attend in-person follow-up data collection events were contacted and offered multiple options for completing the surveys (for example, by web, over the phone, or via mail).

For the implementation evaluation, the evaluation team collected data on attendance, fidelity, and quality. At the end of each module, LiFT facilitators completed an attendance log, a referral log, and a fidelity form. On the fidelity form, they reported whether they covered all of the topics and activities scheduled for that lesson and any deviations from the planned lesson. Trained observers observed more than 10 percent of all sessions to monitor fidelity and quality. The text messaging service recorded the number of text messages sent and received.

ELIGIBILITY:
Inclusion Criteria:

1. Youth must be 13 to 19 years old
2. Youth must live in a rural community that has teen pregnancy rates higher than the national average.
3. Youth must be accompanied by a parenting adult who agrees to participate in the program. The parenting adult does not need to be the youth's biological parent.

Exclusion Criteria:

1. Lack of parental consent
2. Lack of youth assent

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 888 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
No sex or safe sex at last intercourse | 1 year from baseline
  This is a computed dichotomous variable (based on a single survey item - "The last time you had vaginal sex, which of these methods of birth control did you or your partner use?") comprised of youth who reported using any of the following: condom, birth control pills, the shot, the patch, the ring, IUD, implant, or never having vaginal sex as Yes (1) and youth who reported either none, not sure, or other (e.g., withdrawal) as No (0).

SECONDARY OUTCOMES:
No sex or safe sex at last intercourse | 3 months from baseline
  This is a computed dichotomous variable (based on a single survey item - "The last time you had vaginal sex, which of these methods of birth control did you or your partner use?") comprised of youth who reported using any of the following: condom, birth control pills, the shot, the patch, the ring, IUD, implant, or never having vaginal sex as Yes (1) and youth who reported either none, not sure, or other (e.g., withdrawal) as No (0).
Perceived competence in pregnancy prevention scale | 3 months from baseline
  5 survey items having the following responses: strongly agree, agree, disagree, strongly disagree. Items are scored with values 1 to 4, where higher numbers indicate the more favorable response.
  Items that comprise the scale:
  1. If someone asked me where to go for pregnancy prevention methods or other sexual health services, I would know where to send them.
  2. I would feel confident buying condoms or emergency contraception at a drugstore.
  3. If I needed to go to a health clinic for a pregnancy prevention method, I would feel comfortable doing it.
  4. I can use condoms correctly
  5. I can prevent pregnancy easily
  An overall scale score is computed (Alpha=0.8371). The overall scale score is presented on a scale of 0 to 100% based on the percent of the total score possible for the scale.
Parent child communication about sexuality and pregnancy prevention scale | 3 months from baseline
  6 survey items having the following responses: never, once, 2-3 times, 4-5 times, and 6 or more times. Items are scored with values 1 to 5.
  The items included in the scale:
  In the past 3 months, how often have you talked with your parenting adult about each of the following topics?
  1. Your parenting adult(s) values regarding sex and sexuality
  2. Your thoughts and feelings on sex and sexuality
  3. Dating and relationships
  4. Preventing pregnancy and/or STDs and HIV
  5. Consent and saying no to things you don't want sexually
  6. How to use or get condoms or other birth control
  An overall scale score is computed (Alpha=0.8681). The overall scale score is presented on a scale of 0 to 100% based on the percent of the total score possible for the scale.

IPD SHARING:
Plan to Share IPD: No